CLINICAL TRIAL: NCT00515892
Title: A Phase 1, Multicenter, Dose Escalation Study of CAT-8015 in Patients With Relapsed or Refractory Non-Hodgkin'd Lymphoma (NHL)
Brief Title: Safety Study of CAT-8015 Immunoxin in Patients With NHL With Advance Disease
Acronym: NHL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cambridge Antibody Technology (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAT-8015-1003; NCT00522483 (obsolete NCT alias)
Record Dates: First submitted 2007-08-10; First posted 2007-08-14 (Estimated); Last update posted 2007-08-14 (Estimated); Status verified 2007-08

CONDITIONS: Leukemia; Non-Hodgkin's Lymphoma; NHL
MeSH Terms: conditions — Leukemia; Lymphoma, Non-Hodgkin | interventions — immunotoxin HA22; Biological Therapy; Immunization, Passive; Antibodies, Monoclonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Immunotoxin therapy
Drug: CAT-8015 Immunotoxin
Procedure: Biological therapy
Procedure: Antibody Therapy
Procedure: Monoclonal Antibody Therapy

SUMMARY:
RATIONALE: The CAT-8015 immunotoxin can bind tumor cells and kill them without harming normal cells. This may be effective treatment for Non-Hodgkin's lymphoma (NHL) that has not responded to chemotherapy, surgery or radiation therapy.

PURPOSE: Phase 1 dose escalation study to determine the maximum tolerated dose of CAT-8015 immunotoxin in treating patients who have Non-Hodgkin's lymphoma and do not respond to treatment.

ELIGIBILITY:
INCLUSION CRITERIA:

DISEASE CHARACTERISTICS:

* Confirmed diagnosis of B-cell non-Hodgkin's lymphoma
* Measurable disease
* Evidence of CD22-positive malignancy by the following criteria,

  * > 30% of malignant cells from a disease site CD22+ by FACS analysis or,
  * > 15% of malignant cells from a disease site must react with anti-CD22 by immunohistochemistry
* Patients with indolent subtypes of CD22+ B-cell non-Hodgkin's lymphoma, including, but not limited to mantle cell lymphoma, follicular lymphoma and Waldenström's macroglobulinemia, are eligible if stage III-IV.
* Patients must have failed at least two or more courses of prior standard chemotherapy and/or biologic therapy (e.g. Rituxan). Patients with progressive mantle cell lymphoma may be eligible if they have failed one prior standard therapeutic regimen.

PATIENTS CHARACTERISTICS

Performance Status

* ECOG 0-2

Life Expectancy

* Life expectancy of less than 6 months, as assessed by the principal investigator

Other

* Patients with other cancers who meet eligibility criteria and have less than 5 years of disease free survival will be considered on a case-by-case basis
* Must be able to understand and sign informed consent
* Female and male patients must agree to use an approved method of contraception during the study

Exclusion Criteria:

* History of bone marrow transplant
* Documented and ongoing central nervous system involvement with their malignant disease (history of CNS involvement is not an exclusion criterion)
* Pregnant or breast-feeding females
* Patients whose plasma contains either a significant level of antibody to CAT-8015 as measured by ELISA, or antibody that neutralizes the binding of CAT-8015 to CD22 as measured by a competition ELISA.
* HIV positive serology (due to increased risk of severe infection and unknown interaction of CAT-8015 with antiretroviral drugs)
* Hepatitis B surface antigen positive
* Uncontrolled, symptomatic, intercurrent illness including but not limited to: infections requiring systemic antibiotics, congestive heart failure, unstable angina pectoris, cardiac arrhythmia, psychiatric illness, or social situations that would limit compliance with study requirements

Hepatic function: serum transaminases (either ALT or AST) or bilirubin

* ≥ Grade 2, unless bilirubin is due to Gilbert's disease

Renal function: Serum creatinine clearance ≤ 60mL/min as estimated by Cockroft-Gault formula

Hematologic function:

* The ANC < 1000/cmm, or platelet count <50,000/cmm, if these cytopenias are not judged by the investigator to be due to underlying disease (i.e. potentially reversible with anti-neoplastic therapy).
* A patient will not be excluded because of pancytopenia ≥ Grade 3, or erythropoietin dependence, if it is due to disease, based on the results of bone marrow studies
* Baseline coagulopathy > Grade 3 unless due to anticoagulant therapy.

Pulmonary function:

* Patients with < 50% of predicted forced expiratory volume (FEV1) or <50% of predicted diffusing capacity for carbon monoxide (DLCO), corrected for hemoglobin concentration and alveolar volume. Note: Patient with no prior history of pulmonary illness are not required to have PFTs. FEV1 will be assessed after bronchodilator therapy.

Recent prior therapy:

* Cytotoxic chemotherapy, corticosteroids (except stable doses of prednisone), whole body electron beam radiation therapy, hormonal, biologic or other standard or any investigational therapy of the malignancy for 3 weeks prior to entry into the trial
* Less than or equal < 3 months prior monoclonal antibody therapy (i.e. rituximab)
* Patients who are receiving or have received radiation therapy less than 3 weeks prior to study entry will be not be excluded providing the volume of bone marrow treated is less than 10% and also the patient has measurable disease outside the radiation port
* Any history of prior pseudomonas-exotoxin immunotoxin (PE) administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-08

PRIMARY OUTCOMES:
Estimate the maximum dose that can be safely administered to a patient; Characterize the toxicity profile of CAT-8015; Study the clinical pharmacology of CAT-8015; Observe anti-tumor activity, if any.

SECONDARY OUTCOMES:
To assess the immunogenic potential of CAT-8015 to induce antibodies; To investigate the potential of biomarkers to predict any therapeutic or toxic response.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Tower Hematology Oncology Medical Group, Beverly Hills, California
  - Warren Grant Megnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland
- Klinika Hamtologii Uniwersytetu Medycznego (Medical University of Lodz), Lodz, Poland

REFERENCES:
- [Background] Kreitman RJ, Squires DR, Stetler-Stevenson M, Noel P, FitzGerald DJ, Wilson WH, Pastan I. Phase I trial of recombinant immunotoxin RFB4(dsFv)-PE38 (BL22) in patients with B-cell malignancies. J Clin Oncol. 2005 Sep 20;23(27):6719-29. doi: 10.1200/JCO.2005.11.437. Epub 2005 Aug 1. PMID 16061911